

# BIOEQUIVALENCE STUDY PROTOCOL

COMPARATIVE RANDOMIZED, SINGLE DOSE, TWO-WAY CROSSOVER OPEN LABEL STUDY TO DETERMINE THE BIOEQUIVALENCE OF 5 MG/ML TRAMADOL HYDROCHLORIDE ORAL SOLUTION (08P1902F0) RELATIVE TO CONTRAMAL® (100 MG/ML ORAL SOLUTION) AFTER AN ORAL ADMINISTRATION TO HEALTHY ADULTS UNDER FASTING CONDITIONS

Study code: UP-CLI-2021-001 Version 1.0 – 13 February 2022

Sponsor

**UNITHER Pharmaceuticals** 

3-5 Rue Saint-Georges 75009 Paris France



**Test product** 5 mg/mL Tramadol Hydrochloride Oral Solution (08P1902F0)

**Development Phase** Bioequivalence Study

**EudraCT number** 2021-004916-24

CRO:

International Pharmaceutical Research Center (IPRC)



#### CONFIDENTIALITY STATEMENT

The information provided in this document is strictly confidential and is available for review to investigator(s) and appropriate Independent Ethics Committee (IEC) or Institutional Review Board (IRB). It may not be used, reproduced, published or otherwise disclosed without the written authorization from IPRC or the Sponsor.

#### AMENDMENT POLICY

Protocol Amendments are to be written if any procedure in the Protocol needs to be changed. It must be signed by the principal investigator and the Sponsor. Only if all signatures are available, the Protocol Amendment can be considered approved.

Signatures may-where necessary-be submitted by Fax or e-mail. All amendments are to be sent to and approved by the IRB.

The study must not begin or continue before the IRB gives its written approval.



| Sponsor: | UNITHER Pharmaceuticals |
|---|---|
| Address: | 3-5 Rue Saint-Georges, 75009 Paris, France |
| Sponsor's Signatory Representative: | |
| Direct Emergency Phone Number: | Tel.: +33 (0) 1 44 63 51 78 [Droulin Marie-Aline] International Pharmaceutical Research Center (IPRO |
| Contract Research Organization: | |
| Address: | Sport City Circle, Amman, Jordan. |
| Clinical Site: | IPRC Clinical Site |
| Analytical Site: | IPRC Analytical laboratories. |









## IPRC'S PROTOCOL REVISIONS AND APPROVALS





#### SPONSOR'S REPRESENTATIVE PROTOCOL REVISIONS AND APPROVALS



## PRINCIPAL INVESTIGATOR RESPONSIBILITIES

| I, the undersigned, agree: |
|----------------------------|





# TABLE OF CONTENTS

| 1. | INTRODUCTION | 13 |
|---|---|---|
| 1.1. | | |
| 1.2. | Pharmacological properties | 13 |
| 1.3. | Pharmacokinetic properties | 14 |
| 1.4. | Therapeutic indications | 14 |
| 1.5. | Special warnings and precautions for use | |
| 1.6. | Contraindications | 16 |
| 1.7. | | |
| 1.8. | Interaction with other medicinal products and other forms of interaction | 19 |
| 1.9. | Study Medications | 23 |
| 2. | OBJECTIVES | 24 |
| 2.1. | Justification of the study | 24 |
| 2.2. | Risk to benefit ratio | 24 |
| 3. | ETHICS CONSIDERATIONS | |
| 3.1. | Basic Principle | |
| 3.2. | Institutional Review Board (IRB) | |
| 3.3. | | |
| 3.4. | 3 | |
| 3.5. | | |
| 3.6. | | |
| 3.7. | Subjects Compensation | |
| 4. | Investigation | |
| 4.1. | Study Design | |
| 4.2. | Facilities | |
| 4.3. | Laboratory Investigations | |
| 4.4. | | |
| 4.5. | | |
| 4.6. | J | |
| | 4.6.1. Inclusion criteria | |
| | 4.6.2. Exclusion criteria | |
| | METHODS AND PROCEDURES | |
| 5.1. | 0 11 | |
| 5.2. | Subjects Identification | |
| 5.3. | | |
| 5.4. | Method of administration | |
| 5.5. | Product return or destruction | |
| 5.6. | | |
| 5.7. | Study Conduction and Standardization | |
| 5.8.<br>5.9. | 1 0 | |
| | • | |
| | ). Subjects Monitoring | |
| | Biological Samples Handling and Storage | |
| | 2. Case Report Forms | |
| | l. Quality Unit | |
| | 5. Data Quality Assurance | |
| | 5. Audit and on-site Inspection | |
| <b>6.</b> 1. | | |
| 6.2. | • | |
| · · - · | 6.2.1. Adverse events/ serious adverse events/ adverse drug reaction | |
| | 6.2.2. Relationship to the Test Drug | |





| 10. | | OCOL VERSION HISTORY AND SUMMARY OF CHANGES | |
|---|---|---|---|
| 9. | | INCE | |
| 8. | FINAL I | REPORT, SUPPLEMENTARY DOCUMENTATION AND PUBLICATION POLICY | 49 |
| | 7.2.4. | Sample Size Calculation | |
| | <i>7.2.3</i> . | Confidence Intervals and Bioequivalence Evaluation | |
| | 7.2.2. | Analyses of variance (ANOVA) | |
| | 7.2.1. | Descriptive statistics | 47 |
| 7.2. | Statis | tical Analysis | 47 |
| 7.1. | Phari | nacokinetic Analysis | 46 |
| 7. | DATA A | NALYSIS | 46 |
| 6.6. | 6.6. Replacement of withdrawal subjects | | 45 |
| 6.5. | | ct Withdrawal | |
| 6.4. | | fication of the Study Protocol | |
| | | urrent Medications | |
| | 6.2.6. | Follow- up after adverse events | 44 |
| | 6.2.5. | Reporting of adverse events or serious adverse events | |
| | <i>6</i> .2.4. | Subjects' Adverse Events Form | |
| | 6.2.3. | Adverse Event Documentation | 43 |





LIST OF ABBREVIATIONS

ADL Activities of Daily Living
ADR Adverse Drug Reaction

AE Adverse Event

ALP Alkaline Phosphatase ANOVA Analysis Of Variance

ATC Anatomic Therapeutic Chemical classification
AUC Area Under the plasma concentration-time Curve

 $AUC_{0\rightarrow t}$  Area Under the plasma concentration-time Curve from zero

(0) hours to time (t) hours

AUC<sub> $0\to\infty$ </sub> Area Under the plasma concentration-time Curve from zero (0) hours to

infinity  $(\infty)$ 

BMI Body Mass Index BUN Blood Urea Nitrogen

°C Celsius cm Centimeter

C<sub>max</sub> Maximal Plasma Concentration.

CNS Central Nervous System
COVID-19 Corona virus Disease 2019

CRF Case Report Form.

CRO Contract Research Organization

CYP Cytochrome P.
CV Curriculum Vitae
DMU Data Management Unit
ECG Electrocardiogram

EMA European Medicines Agency

g Gram

GCP Good Clinical Practice
GLP Good Laboratory Practice
GMP Good manufacturing practice

Hr/h Hour

HBsAg Hepatitis B surface Antigen HCG Human chorionic gonadotropin

HCl Hydrochloride

HIV Human Immunodeficiency Virus

ICF Informed Consent Form.

ICH International Council for Harmonization

IEC Independent Ethic Committee
IMP Investigational Medicinal Product

IPRC International Pharmaceutical Research Center

IRB Institutional Review Board
ISR Incurred Sample Reanalysis





# LIST OF ABBREVIATIONS (CONTINUED)

JFDA Jordan Food and Drug Administration

K<sub>el</sub> Elimination rate constant.

Kg Kilogram
L Liter
Log Logarithm

LogP log partition coefficient

LLOQ Lower Limit of Quantification

m<sup>2</sup> meter square

MAOIs Monoamine Oxidase Inhibitors MCV Mean corpuscular volume

MCH Mean Corpuscular Haemoglobin

MCHC Mean Corpuscular Haemoglobin -Concentration

mg milligram minutes mL milliliter

mmHg millimeter of mercury PCV Packed cell volume

pH Measure of the acidity or basicity of a solution.

PKa Negative log of the acid dissociation constant or Ka value QTc is a measure of the time between the start of the Q wave and

the end of the T wave in the heart's electrical cycle.

QU Quality Unit

SAE Serious Adverse Events

SGOT (AST) Serum Glutamic Oxalate Transaminase (Aspartate

Aminotransferase)

SGPT (ALT) Serum Glutamic Pyruvate Transaminase (Alanine

Transaminase)

SmPC Summary of Product Characteristics

SNRIs Serotonin and Norepinephrine Reuptake Inhibitors

SOP Standard Operating Procedure

SSRIs Selective Serotonin Reuptake Inhibitors

 $t_{1/2el}$  Half Life

t<sub>max</sub> Time point of maximal plasma concentration





# SUMMARY OF MAJOR STUDY DATA

| | SUMMARY OF MAJOR STUDY DATA |
|---|---|
| TITLE | Comparative Randomized, Single Dose, Two-Way Crossover Open Label Study To Determine The Bioequivalence Of 5 mg/mL Tramadol Hydrochloride Oral Solution (08P1902F0) Relative To Contramal® (100 mg/mL Oral Solution) After An Oral Administration To Healthy Adults Under Fasting Conditions |
| OBJECTIVES | <b>Primary Objective:</b> The aim of this study is to determine the bioequivalence between Test Product relative and Reference Product in terms of AUC (Area under the curve) and C <sub>max</sub> after a single oral dose administration of 50 mg tramadol hydrochloride to healthy adults under fasting conditions <b>Secondary Objective:</b> To investigate the safety and tolerability of the formulations. |
| STUDY ETHICAL | The study will be conducted according to the "Declaration of Helsinki". |
| CONDUCTION | 8 |
| STUDY DESIGN | Screening period Wash-out 2 1 week Cross-Over To T24h To T24h To T24h Somg (10mL) 08P1902F0 (tramadol hydrochloride, oral solution 5mg/mL) B 50mg (0,5mL = 20 drops) of Contramal® (tramadol hydrochloride oral solution 100mg/mL) |
| STUDY SUBJECTS | Healthy male or female subjects, 18-50 years of age, selected from the Jordan population and fulfilling the selection criteria. 24 male or female subjects plus 1-2 alternates will be admitted to the study. |
| Dosage Regimen | A single oral dose of 50 mg tramadol hydrochloride oral solution from each product will be administered according to a randomization scheme. |
| ADMISSION AND<br>CONFINEMENT | Subjects will be admitted the night before the study drug administration, supervised for at least 10 hours of overnight fasting, and confined until collecting the 24-hour sample. |
| ANCILLARY<br>ASSESSMENT | Safety/adverse events, laboratory evaluation, ECG, physical examination, vital signs and evaluation of palatability. |





SUMMARY OF MAJOR STUDY DATA (CONTINUED) Eighteen blood samples will be collected in lithium heparinized tubes before dosing BLOOD SAMPLING Drug assays will be carried out using validated chromatographic methods developed specifically for the determination of tramadol in plasma using an achiral BIOANALYSIS assay and its active metabolite O-desmethyltramadol in plasma Primary Pharmacokinetic Parameters of tramadol: C<sub>max</sub> and AUC<sub>0→t</sub>. **PHARMACOKINETICS** AND STATISTICAL ANALYSIS The confidence intervals of logarithmically transformed Test/Reference ratios for  $C_{\text{max}}$  and  $AUC_{0\rightarrow t}$  are set to be within 80.00-125.00%. BIOEQUIVALENCE CRITERIA FINAL REPORT A comprehensive report will be issued after completion the study.





# 1. Introduction

# 1.1. Chemistry<sup>1</sup>

Tramadol hydrochloride is an opioid agonist. The chemical name for tramadol hydrochloride is (±)cis-2- [(dimethylamino)methyl]-1-(3-methoxyphenyl) cyclohexanol hydrochloride. The structural formula is:

The molecular formula of tramadol hydrochloride is  $C_{16}H_{25}NO_2 \cdot HCl$ , and the molecular weight is 299.8. Tramadol hydrochloride is a white, bitter, crystalline and odorless powder. It is readily soluble in water and ethanol and has a pKa of 9.41. The n-octanol/ water log partition coefficient (logP) is 1.35 at pH 7. Tramadol hydrochloride oral solution (08P1902F0) is a clear, raspberry cherry flavored liquid containing 5 mg of tramadol hydrochloride per 1 mL (equivalent to tramadol 4.4 mg per 1 mL)

# 1.2. Pharmacological properties<sup>2</sup>

## Pharmacotherapeutic group: other opioids; ATC-code: N 02 AX02. Class

Tramadol is a centrally-acting opioid analgesic. It is a non-selective pure agonist at  $\mu$ ,  $\delta$  and  $\kappa$  opioid receptors with a higher affinity for the  $\mu$  receptor. Other mechanisms which contribute to its analgesic effect are inhibition of neuronal re-uptake of noradrenaline and enhancement of serotonin release.

Tramadol has also an antitussive effect. In contrast to morphine, analgesic doses of tramadol over a wide range have no respiratory-depressant effect. Also gastrointestinal motility is less affected. Effects on the cardiovascular system tend to be slight.

The potency of tramadol is reported to be 1/10 (one tenth) to 1/6 (one sixth) that of morphine.





# 1.3. Pharmacokinetic properties<sup>2</sup>

#### In adults

After a single oral administration of a dose of 50 to 100 mg, the bioavailability is between 70 and 90%.

After oral administration, repeated every 6 hours, of 50 to 100 mg, the state of equilibrium is quickly reached in about 36 hours and the bioavailability increases, exceeding 90%.

The peak serum after oral administration of 100 mg of tramadol is approximately 300 ng / mL ( $C_{max}$ ) and is reached after approximately 2 h ( $t_{max}$ ).

Plasma protein binding is 20%, and the volume of distribution is large (3 to 4 l/kg). Tramadol crosses the placental barrier and passes in very small amounts into breast milk (approximately 0.1% of the maternal dose administered).

Elimination half-life is between 5 and 7 hours in healthy volunteers; 90% of tramadol is metabolized, mainly in the liver; one of the demethylated metabolites has an analgesic effect; its half-life is of the same order as that of tramadol.

Tramadol and its metabolites are almost completely excreted via the kidneys (95%). The rest is eliminated in the faeces.

The pharmacokinetics of tramadol are only slightly affected by the age of the patient.

In patients with renal impairment, the clearance of tramadol is reduced in parallel with the clearance of creatinine; the half-life is on average 12 hours.

In hepatic impairment, the clearance of tramadol is reduced, depending on the severity of the hepatic impairment.

# 1.4. Therapeutic indications<sup>2</sup>

Treatment of moderate to severe pain.





1.5. Special warnings and precautions for use as indicated in SmPC of Contramal®. Some of them are not applicable to the protocol (single dose, adult healthy population, exclusion criteria ect...)<sup>2</sup>

# Special warnings

# Children and rapid metabolizer

- Those close to the child should be informed that this oral solution should be kept out of reach of children (locked up) to avoid any risk of accidental overdose which could have potentially fatal consequences.
- Cases of ultra-rapid metabolizers have been reported, especially in children.
- Parents should be informed, especially during the first administration, of the need to
  monitor their child, and to call a doctor or emergency service in case of any unusual signs,
  including disturbances of consciousness, miosis, vomiting, convulsions or respiratory
  depression.

# Other warnings

Tramadol should be used with particular caution in opioid-dependent patients, in patients predisposed to seizures or in patients with head injury, shock, a reduced level of consciousness of uncertain origin, disorders of the respiratory center or function, increased intracranial pressure.

In opioid dependent patients and in patients with a history of abuse or dependence, treatment should be short-term and under strict medical supervision.

Tramadol is not suitable for substitution therapy in patients with opioid dependence. Although an opioid agonist, tramadol cannot correct the symptoms of opioid withdrawal.

Tolerance and physical and / or psychological dependence can develop even at therapeutic doses. The clinical need for analgesic treatment should be reviewed regularly.

Cases of dependence and abuse have been reported.

Withdrawal symptoms, similar to those which occur with opioid withdrawal, could occur. Withdrawal symptoms can be avoided by gradually reducing the dose when stopping treatment, especially after long periods of treatment.





Special care should be taken when treating patients with respiratory depression or if concomitant CNS depressant drugs are being administered, or if the recommended dosage is significantly exceeded, as the possibility of respiratory depression cannot be excluded in these situations.

Concomitant use of Tramadol with morphine agonist-antagonists (buprenorphine, nalbuphine, pentazocine), and carbamazepine is not recommended.

Alcohol intake during treatment is not recommended.

Convulsions have been reported in patients receiving tramadol at the recommended dose levels. The risk may be increased when doses of tramadol hydrochloride exceed the recommended upper daily dose limit (400 mg). In addition, tramadol may increase the seizure risk in patients taking other medicinal products that lowers the seizure threshold. Patients with epilepsy or those susceptible to seizures should only be treated with tramadol if there are compelling circumstances.

This medicine contains castor oil and may cause digestive problems (mild laxative effect, diarrhea).

This medicine contains a derivative of sucrose. Its use is not recommended in patients with fructose intolerance, glucose-galactose malabsorption syndrome or sucrase-isomaltase deficiency.

# Precautions for use

Tramadol should only be used after careful assessment of the risk-benefit ratio, depending on the origin of the pain and the profile of the patient.

#### 1.6. Contraindications<sup>2</sup>

Tramadol is contraindicated

- In hypersensitivity to the active substance or any of the excipients;
- In acute intoxication with alcohol, hypnotics, analgesics, opioids or other psychotropic medicinal products;
- In patients who are receiving MAO inhibitors, especially with linezolid, and methylene blue or who have taken them within the last 14 days;
- In case of severe respiratory failure;





- In children under 3 years old;
- in patients with epilepsy not adequately controlled by treatment;
- for use in narcotic withdrawal treatment.

This medicine should generally not be used:

during pregnancy.

#### 1.7. Adverse Events<sup>2</sup>

The most commonly reported adverse reactions are nausea and dizziness, both occurring in more than 10 % of patients.

The frequencies are defined as follows:

Very common:  $\geq 1/10$ 

Common:  $\geq 1/100$ , < 1/10

Uncommon: >1/1000, <1/100

Rare:  $\geq 1/10~000$ , < 1/1000

Very rare: <1/10 000

Not known: cannot be estimated from the available data

#### **Immune system disorders:**

• Rare: allergic reaction (eg., dyspnea, bronchospasm, wheezing, angioedema) and anaphylaxis.

## **Psychiatric disorders:**

• <u>Rare:</u> hallucinations, confusion, sleep disturbance, delirium, anxiety, nightmares. After administration of tramadol, various psychological side effects may also be observed, the intensity and nature of which vary from one patient to another (depending on the individual reactivity and the duration of the treatment.). changes in mood (usually elation, occasionally dysphoria), changes in activity (usually decreased activity, occasionally increased), and changes in cognitive and sensory abilities (for example, decision behaviour, perception disorders).

Cases of abuse and dependence have been reported as well as cases of withdrawal syndrome.

Withdrawal symptoms, similar to those seen during opioid withdrawal, may occur such as restlessness, anxiety, nervousness, insomnia, hyperkinesia, tremors, and gastrointestinal symptoms.





Other withdrawal symptoms have been reported very rarely, including: panic attack, severe anxiety, hallucinations, paraesthesia, tinnitus, other CNS disorders (eg confusion, delirium, depersonalization, derealization, paranoia).

# Nervous system disorders:

- Very common: Dizziness
- <u>Common</u>: Headache, somnolence
- <u>Rare</u>: paraesthesia, tremor, convulsions, involuntary muscle contractions, abnormal coordination, syncope, Speech disorders

Convulsion have mainly occurred after administration of high doses of tramadol or after concomitant treatment with drugs which may lower the seizure threshold.

• <u>Unknown</u>: loss of consciousness.

# Metabolism and nutrition disorders

- Rare: change in appetite.
- *Unknown*: hypoglycemia

# Eye disorders:

• Rare: miosis, blurred vision, mydriasis.

# Cardiovascular disorders:

- <u>Uncommon</u>: effects on cardiovascular regulation (palpitation, tachycardia). These side effects may occur especially after intravenous administration and in patients under physical stress.
- Rare: bradycardia

#### Vascular disorders:

• <u>Uncommon</u>: effects on cardiovascular regulation (orthostatic arterial hypotension or cardiovascular collapse). These side effects may occur especially after intravenous administration and in patients under physical stress.

# Respiratory, thoracic and mediastinal disorders:

• Rare: respiratory depression, dyspnea.

Respiratory depression may occur if the doses administered greatly exceed the recommended doses and if other central depressant drugs are administered concomitantly.

Worsening asthma has also been reported, although a causal relationship has not been established.





# **Gastrointestinal disorders:**

- · Very common: nausea.
- Common: Constipation, dry mouth, vomiting.
- <u>Uncommon</u>: retching, gastrointestinal irritation (a feeling of pressure in the stomach, bloating), diarrhoea.

# Hepatobiliary disorders

• In a few isolated cases an increase in liver enzymes has been reported with the therapeutic use of tramadol.

## Skin and subcutaneous tissue disorders

- · Common: sweating
- Uncommon: Dermal reactions (Pruritus, rash, urticaria)

# Musculo-skeletal disorders:

• Rare: Motorial weakness

# Renal and urinary disorders

• Rare: Micturition disorders (dysuria and urinary retention)

## General disorders and administration site conditions

· Common: asthenia

# **Investigations**

• *Rare*: increase in blood pressure

# 1.8. Interaction with other medicinal products and other forms of interaction<sup>2</sup>

The results of pharmacokinetic studies have so far shown that on the concomitant or previous administration of cimetidine (enzyme inhibitor) clinically relevant interactions are unlikely to occur.

# **Drugs causing serotonin syndrome**

Tramadol can induce convulsions and increase the potential for selective serotonin re-uptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, anti-psychotics and other seizure threshold-lowering medicinal products (such as bupropion, mirtazapine, tetrahydrocannabinol) to cause convulsions.





Concomitant therapeutic use of tramadol and serotonergic drugs, such as selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), MAO inhibitors, tricyclic antidepressants and mirtazapine may cause serotonin toxicity: diarrhea, tachycardia, sweating, tremors, confusion or even coma

Withdrawal of the serotoninergic medicinal products usually brings about a rapid improvement. Treatment depends on the type and severity of the symptoms.

Other active substances known to inhibit CYP3A4, such as ketoconazole and erythromycin, might inhibit the metabolism of tramadol (N-demethylation) probably also the metabolism of the active O-demethylated metabolite. The clinical importance of such an interaction has not been studied.

# Drugs lowering the seizure threshold

The concomitant use of proconvulsant drugs, or drugs lowering the epileptogenic threshold, should be carefully weighed, due to the severity of the risk involved. These drugs are represented in particular by most antidepressants (imipramines, selective serotonin reuptake inhibitors), neuroleptics (phenothiazines and butyrophenones), mefloquine, chloroquine, bupropion, fluoroquinolones, tramadol.

# Sedative drugs

It should be taken into account that many drugs or substances can add up their depressant effects on the central nervous system and contribute to reducing vigilance. These are morphine derivatives (analgesics, cough suppressants and substitution treatments), neuroleptics, barbiturates, benzodiazepines, anxiolytics other than benzodiazepines (for example, meprobamate), hypnotics, sedative antidepressants (amitriptyline, doxepine, mianserin, mirtazapine, trimipramine), sedating H1 antihistamines, central antihypertensive drugs, baclofen and thalidomide.

# **Contraindicated combinations**

#### + Irreversible MAOIs (iproniazid)

Risk of the appearance of a serotonin syndrome: diarrhea, tachycardia, sweating, tremors, confusion or even coma.

Allow two weeks between stopping MAOI and starting treatment with tramadol, and at least one week between stopping tramadol and starting MAOI.





# Not recommended associations

# + Morphinic agonists-antagonists (buprenorphine, nalbuphine, pentazocine)

Decrease in the analgesic effect by competitive blocking of receptors, with the risk of the appearance of a withdrawal syndrome.

# + Alcohol (drink or excipient)

Alcohol enhancement of the sedative effect of morphine analgesics.

Impaired alertness can make driving and using machines dangerous.

Avoid taking alcoholic drinks and drugs containing alcohol.

#### + Carbamazepine

Risk of decreased plasma concentrations of tramadol.

Co-administration or prior administration of carbamazepine (enzyme inducer) may reduce analgesic effects and shorten the duration of action of tramadol.

# + Reversible MAOIs including linezolid and methylene blue

Risk of the appearance of a serotonin syndrome: diarrhea, tachycardia, sweating, tremors, confusion or even coma.

If the combination cannot be avoided, very close clinical monitoring. Start the combination at the minimum recommended doses.

## + Partial antagonist morphines

Risk of reduction of the analgesic effect.

#### + Naltrexone

Risk of reduction of the analgesic effect.

## + Sodium oxybate

Increase in central depression

Impaired alertness can make driving and using machines dangerous.





# Combinations subject to precautions for use

#### + Antivitamin K

Risk of increased effect of antivitamin K and risk of bleeding. More frequent monitoring of the INR. Possible adjustment of the dose of the antivitamin K during treatment with tramadol and after its discontinuation.

# Associations to take into account

+ Other opioid agonist analgesics, morphine-like cough suppressants (dextromethorphan, noscapine, pholcodine), true morphine cough suppressants (codeine, ethylmorphine)

Increased risk of respiratory depression which may be fatal in case of overdose.

# + Other drugs lowering the seizure threshold

Increased risk of convulsion.

## + Other sedative drugs

Increase in central depression.

Impaired alertness can make driving and using machines dangerous.

# + Benzodiazepines and related drugs

Increased risk of respiratory depression which may be fatal in case of overdose.

#### + Barbiturates

Increased risk of respiratory depression which may be fatal in case of overdose.

#### + MAOI B

Risk of onset of serotonin syndrome.

# + Selective serotonin reuptake inhibitors (citalopram, escitalopram, fluoxetine, fluoxetine, paroxetine, sertraline)

Risk of onset of seizures and / or serotonin syndrome.

#### + Venlafaxine

Risk of onset of seizures and / or serotonin syndrome.





# + Buproprion

Increase in plasma concentrations of tramadol due to decrease in its hepatic metabolism by bupropion. In addition, risk of seizures due to the addition of the effects of the two drugs.

## + Ondansetron

Decreased strength and duration of analgesic effect of tramadol and risk of reduced antiemetic effect of ondansetron.

# 1.9. Study Medications

| Identification | TEST Product -Treatment A | REFERENCE Product-Treatment B |
|----------------|---------------------------|-------------------------------|
| | | /-2 mL of water |





# 2. OBJECTIVES

**Primary Objective:** This aim of this study is to demonstrate the bioequivalence between Test Product and Reference Product after a single oral dose administration of 50 mg tramadol hydrochloride to healthy adults under fasting conditions. The bioequivalence of a single dose of 50 mg tramadol hydrochloride will be assessed by comparing the pharmacokinetic parameters derived from the plasma concentration-time profiles of tramadol.

**Secondary Objective:** To investigate the safety and tolerability of the formulations.







| Ī |
|---|
| i |
| ı |





## 3. ETHICS CONSIDERATIONS

#### 3.1. Basic Principle

This research will be carried out in accordance with conditions stipulated by International clinical research guidelines and the principles enunciated in the Declaration of Helsinki<sup>3</sup> and the ICH harmonized tripartite guideline regarding Good Clinical Practice (GCP) adopted by the European Medicines Agency<sup>4</sup> guidelines for bioequivalence. In addition, all local regulatory requirements will be adhered to, in particular those which afford greater protection to the safety of the study participants<sup>5</sup>.

## 3.2. Institutional Review Board (IRB)

The Institutional Review Board of the IPRC will review the protocol and the study will not start until the Board has approved the protocol or a modification thereof. The Board is constituted and operates in accordance with the principles and requirements described in the Guidelines on Research Involving Human Subjects<sup>6</sup>. All amendments to the study protocol are to be sent to the IRB for approval.

## 3.3. Informed Consent

The purpose of the study, the procedures to be carried out and the potential hazards will be described to the subjects in non-technical terms. Subjects will be required to read, sign and date a consent form summarizing the discussion prior to enrolment and will be assured that they may withdraw from the study at any time without jeopardizing their medical care. IPRC will keep the ICF for the subjects also a copy will be given to the subject.

# 3.4. Subject Confidentiality

All communications and documents relevant to subjects in the study will identify each subject only by the subjects' initials or by the subjects' study numbers.

# 3.5. Study Completion, Termination or Suspension

The Principal Investigator will complete this study in satisfactory compliance with the study protocol. It is agreed that, for a reasonable cause, either the Principal Investigator, JFDA, IRB or Sponsor may terminate this study prematurely, provided that written notice is submitted at a reasonable time in advance of the intended termination.







| insurance company. Each subje | ct will be informed | about his indemnit | y in the Informed | l Consent |
|---|---|---|---|---|
| | l | | | |





#### 4. Investigation

# 4.1. Study Design<sup>7,8</sup>

Open-label, randomized, two-way crossover study to compare the relative bioavailability of tramadol from Test product and Reference Product given as a single dose of 50 mg tramadol hydrochloride under fasting conditions. The subjects who conform to the study entry criteria will be dosed according to a randomization schedule. The plan of study is depicted in Figure 1.

Figure 1 Study Plan



#### 4.2. Facilities

The clinical part of the study will be performed at the IPRC clinical site, a clinical site with examination rooms; procedural laboratories and emergency care equipment. Drug assays will be performed at the IPRC analytical laboratories. Pharmacokinetics and biostatistical analysis will be performed by the data management unit. All facilities are located in Amman, Jordan.





# 4.3. Laboratory Investigations

Before enrolment in the study, the subjects will undergo clinical laboratory tests performed by the IPRC clinical laboratories.

# 4.4. Screening and follow up



In case of withdrawals, if the subject received the study's medication at least once, follow-up examinations will be done according to the nature of the withdrawal. If the subject withdraws because of adverse event(s), the Principal Investigator will arrange close monitoring of the subject with the necessary measurements. Subject who have an acute infection within one week preceding study drug administration will not be admitted to the study.





Table 1 Laboratory tests to be performed on subjects.

| Tests | Screening | Before<br>admission<br>to period I | Before<br>admission<br>to period II | Follow Up |
|---|---|---|---|---|
| | Haen | natology | | |
| | | | | _ |





# 4.5. Study Subjects

24 male or female subjects plus 1-2 alternates will be admitted in the study.

# 4.6. Subject Selection Criteria

To be eligible for participation in the study, subjects must meet all of the following criteria before their enrolment in the study.

# 4.6.1. Inclusion criteria

- 1. Healthy subjects male or female, age 18 to 50 years, inclusive.
- 2. Body weight  $\geq$  50 kg.
- 3. Body Mass Index (BMI) range<sup>8</sup> is within  $18.5 30 \text{ Kg/m}^2$ .







#### 4.6.2. Exclusion criteria

- 1. Medical history performed not longer than two weeks before the initiation of the clinical study with significant deviations from the normal ranges.
- 2. Presence of any clinically significant results from laboratory tests, however, ALP and creatinine will be accepted if below the reference range after being evaluated by the physician as clinically not significant. Haematology tests with deviation of more than 5% of the reference limits. Laboratory tests are performed not longer than two weeks before the initiation of the clinical study.













# 5. METHODS AND PROCEDURES

# 5.1. Drug Supplies and Retention

| The Sponsor will supply sufficient quantities of the study Investigational Medicinal Products to |
|---|
| allow completion of this study. |
| 5.2. Subjects Identification |
| 5.3. Randomization |
| 5.4. Method of administration |
| Only subjects enrolled in the study may receive investigational product, in accordance with all applicable regulatory requirements. Only authorized site staff may supply or administe investigational product. |





#### 5.5. Product return or destruction

At the end of the study, there will be a final reconciliation of product shipped, product consumed, product remaining and treatment disposed. This reconciliation will be recorded in the accountability record form, signed and dated.

Remaining IMP will either be disposed at the study site according to the study site's institutional standard operating procedure or be returned to Creapharm with the appropriate documentation. The site's method of destroying Sponsor-supplied IMPs must be agreed by the Sponsor. The site must obtain written authorization from the Sponsor before any Sponsor-supplied IMP is destroyed, and IMP destruction must be documented on the appropriate form.

Any discrepancies noted will be investigated, resolved and documented prior to destruction.

#### 5.6. Restrictions and Prohibitions









# 5.7. Study Conduction and Standardization

Subjects will only be included in the study, if they participate in a meeting with the Principal Investigator or the clinical staff about the details of the study, if they give their written informed consent, if they meet the inclusion criteria and do not meet the exclusion criteria, and if the Principal Investigator gives the final approval for the subjects to participate after completion of the screening part. The study is to be conducted as proposed below:

• In the evening before administration on study day 1 of study periods I and II, subjects will be admitted to the clinical site.












# 5.9. End of study

The end-of-study is defined as the date of the last subject's last assessment.

# 5.10. Subjects Monitoring



## 5.11. Biological Samples Handling and Storage

Blood samples will be collected at the times specified under the sampling schedule, and centrifuged (using refrigerated centrifuge) as soon as possible after collection. Following centrifugation, the resulting plasma will be transferred directly into plain plastic tubes. These samples will be stored at the clinical site at around -70°C using dry ice till transferred to the freezers area to be stored in the -70°C freezers. All plasma samples will be divided into two (2) aliquots. All samples will be collected into suitably labelled tubes (subject no., part one from study code, the year the study was assigned and the number of the study, study period, sample no. and aliquot no.).





# 5.12. Case Report Forms

The IPRC will supply Case Report Forms (CRFs). Case Report Forms must be completed for each subject enrolled in this study and will be reviewed at the end of each study period for completeness and acceptability by IPRC personnel at the study site.

# 5.13. Drug Bioanalysis







## 5.14. Quality Unit

The Quality Unit (QU) of IPRC will be responsible for the conduction of the study according to the GLP, ICH-GCP guidelines, the most recent revised version of the Declaration of Helsinki (Fortaleza, October 2013), the applicable regulatory requirement, the study protocol and the inhouse SOP's, for both the clinical and analytical tasks. A complete audit is to be performed by the QU for the overall study execution. A final quality unit statement will be issued to indicate each audit task.

## 5.15. Data Quality Assurance

Monitoring details describing strategy, methods, responsibilities and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the Monitoring Plan.

Study monitor, designated by Sponsor will perform source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of patients are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all local applicable regulatory requirements.

Records and documents, including signed ICFs, pertaining to the conduct of this study must be retained by the investigator for 25 years after study completion unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the Sponsor. No records may be transferred to another location or party without written notification to the Sponsor.

## 5.16. Audit and on-site Inspection

Prior to the start of the study, the investigator is required to confirm his/her agreement to conduct the study in accordance with the protocol and to give access to all relevant data and records to UNITHER Pharmaceuticals monitors, auditors, and designated agents of UNITHER Pharmaceuticals, IRBs/IECs, and regulatory authorities as required.

If an inspection of the site is requested by a regulatory authority for this study, the investigator must inform UNITHER Pharmaceuticals and designated agents of UNITHER Pharmaceuticals (Monitor) immediately that this request has been made.





## 6. Management of Intercurrent Events

## 6.1. Deviation from Study Protocol for the individual subject

When significant deviation from the Study Protocol is deemed necessary for an individual subject, the Principal Investigator or any person assigned by him must contact the Sponsor. Such contact with the Sponsor will be made as soon as possible to permit a decision as to whether or not the subject is to continue in the study. Any deviation from the Study Protocol will be authorized only for that one subject. A description of the deviation from the Clinical and the reason(s) for it will be recorded on the appropriate Case Report Form.

#### 6.2. Adverse Events

Subjects will be monitored throughout confinement for adverse events to the study formulations and/or procedures. The Study Physician or a medically qualified designee will be on site till the end of confinement and on call for the end of the study. At the time of the last blood collection in each study period, each subject will be asked how he/she is feeling. The Study physician will evaluate the situation and take any necessary action. At the beginning of the second period, subjects will be questioned concerning unusual symptoms, which may have occurred after the previous administration of the study drug. The Study Physician or a qualified medical designee will evaluate drug-related symptoms of clinical significance before the next dose is administered. All adverse events and treatment administered will be recorded in the final report.

# 6.2.1. Adverse events/ serious adverse events/ adverse drug reaction<sup>11</sup>

- Adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), for example, symptom or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product.
- Serious Adverse Event (SAE) is one that suggests a significant hazard, contraindication, side effect, or precaution. A serious adverse drug event includes any event that:
  - -Results in death
  - -Is life threatening
  - -Requires patient hospitalization or prolongation of existing hospitalization.
  - -Results in persistent or significant disability / incapacity (as per reporter's opinion)
  - Is a congenital anomaly / birth defect.
  - -Or other seriousness beyond common definitions such as important medical events which might jeopardize the patient or require intervention to prevent the other outcomes as listed in other definitions of seriousness.





 Adverse Drug Reaction (ADR) is a response to a drug which is noxious and unintended, that occurs at doses normally used in man for prophylaxis, diagnosis, modification of a physiological function or therapy of a disease.

The Study Physician will determine in the course of the study whether any adverse events have occurred and will rate their intensity as follows:

Mild: asymptomatic or mild symptoms; clinical or diagnostic

observations only; no intervention indicated

Moderate: minimal, local or non-invasive intervention indicated; limiting age-

appropriate instrumental ADL

Severe or medically significant but not immediately life threatening: hospitalization

or prolongation of hospitalization indicated; disabling; limiting self

care ADL

Life-threatening consequences: urgent intervention indicated

Death related to AE.

# 6.2.2. Relationship to the Test Drug

The Principal Investigator will judge whether or not, in his opinion, the adverse drug reaction was related with the drug. The study physician will decide if the adverse event is drug-related or not related. Nevertheless, the adverse event is to be recorded as follows:

Certain/related: A clinical event, including laboratory test abnormality,

occurring in a plausible time relationship to drug administration and which concurrent disease or other drugs

or chemicals cannot explain.

Probable/likely: A clinical event, including laboratory test abnormality, with

a reasonable time sequence to administration of the drug, unlikely to be attributed to concurrent disease or other drugs or chemicals and which follows a reasonable response on

withdrawal (dechallenge).

Possible: A clinical event, including laboratory test abnormality, with

a reasonable time sequence to administration of the drug, but which could also be explained by concurrent disease or other drugs or chemicals. Information on drug withdrawal may be

lacking or unclear.

Unlikely: A clinical event, including laboratory test abnormality with

a temporal relationship to drug administration which makes a causal relationship improbable and in which other drugs,





chemicals or underlying disease provide plausible

explanation.

Unrelated: A clinical event, including laboratory test abnormality,

which can be explained by any reason excluding the

administered drug.

Not assessable/unclassified: A report suggesting an adverse event that cannot be judged

because information is insufficient or contradictory and

which cannot be supplemented or verified.

### 6.2.3. Adverse Event Documentation

The recording of every AE/ SAE has to meet the following requirement:

- -Subject identification number and initials.
- -Exact documentation of the event.
- -Exact description of temporary sequence to the therapy course when experienced.
- -Documentation of severity.
- -Documentation of the results of diagnostic and therapeutic measurements.
- -Results of repeated exposure if possible.
- -Details of the development and outcome including medical assessment
- -As much data as possible must be obtained which are important for the assessment concerning the relationship of the AE/SAE to study drug.
- -Critical examination of the relationship to study drug.

## 6.2.4. Subjects' Adverse Events Form

Subject will be given an Adverse Events Form (in Arabic language) on Day 1 of each Study Period. Subjects will be asked for side effects, or unexpected events. Separate form will be used for each study period.

## 6.2.5. Reporting of adverse events or serious adverse events







# 6.2.6. Follow- up after adverse events

All adverse events and serious adverse events must be followed up until a conclusion is reached. Any subject withdrawn from the study due to any adverse event will be followed up until a conclusion is reached, also. This conclusion must be reported in the CRFs and to the Sponsor, in the event of an SAE.

#### 6.3. Concurrent Medications



## 6.4. Modification of the Study Protocol

Neither the Principal Investigator, nor the Sponsor will modify this Study Protocol without first obtaining the concurrence of others. The modification must be documented in writing and signed by the Principal Investigator and the Sponsor. Any change in research activity, except for those necessary to remove an apparent immediate hazard to a subject, must be reviewed and approved by the IRB before implementation.

# 6.5. Subject Withdrawal

Each subject has the right to withdraw from the study at any time without jeopardy or prejudice. The Principal Investigator or the Study Physician may discontinue any subjects' participation when he feels it is necessary for any reason including adverse events or failure to comply with the study protocol. Should a subject withdraw from the study, the reasons must be stated on the Case Report Form and a final evaluation of the subject will be performed.





When a subject withdraws after having received the dose, he/she has to be informed by the principal investigator when he/she can take drugs again. This may become especially important when the subject withdraws for medical reasons, which may require drug therapy.

Furthermore, participation in this clinical study could be discontinued by the Principal Investigator or by the Sponsor for any of the following reasons:

- Adverse events;
- Significant protocol violation such as restrictions regarding alcohol and drug use, and non-respect of the fasting conditions;
- Difficulties with blood collection;
- Emesis following drug administration (subjects who experience emesis during the course
  of a bioequivalence study for immediate-release products, should be deleted from
  statistical analysis if vomiting occurs at or before 2 times median t<sub>max</sub>).

The Principal Investigator can also remove a subject from the study if it is determined that the subject is uncooperative during the study. The Principal Investigator can remove a subject from the study due to an unanticipated event that could result in an inadequately characterized profile, such as missed blood draws, an adverse event such as diarrhea or a meal deviation. Details of reasons for removal of subjects will be recorded, reported to the Sponsor and documented in the final report.

## 6.6. Replacement of withdrawal subjects

If a subject is withdrawn before the first study drug administration, he/she will be replaced by the next qualifying alternate. The replacing alternate subject will receive the study products in the same sequence and under the same conditions as the dropped subject, and he/she will undergo the entire protocol procedure. Withdrawals after study drug administration will not be replaced.

When a subject is withdrawn from the study, the reasons are stated on the Case Report Form and a final evaluation of the subject will be performed.





## 7. DATA ANALYSIS

# 7.1. Pharmacokinetic Analysis 12,13







# 7.2. Statistical Analysis 14,15

Samples from all subjects who complete the study will be analyzed for the plasma concentrations and considered for statistical analysis. Samples from withdrawals, if any, will be analyzed if the profile of at least one period can be determined. If necessary, an unequal number of subjects per sequence will be used.

The pharmacokinetic results from withdrawals who do not provide evaluable data for both the test and reference products will not be included in statistical evaluation. Concentration data and pharmacokinetic parameters from such subjects will be presented in the individual listings but will not be included in the summary statistics.



## 7.2.1. Descriptive statistics

Descriptive statistics, including the means, standard deviations, standard error of the mean and coefficient of variation, shall be reported for the plasma concentrations. For pharmacokinetic parameters, arithmetic means, standard deviations, standard error of the mean, minimum, median, maximum, coefficient of variation and geometric mean shall be reported.







7.2.3. Confidence Intervals and Bioequivalence Evaluation



7.2.4. Sample Size Calculation





## 8. Final Report, Supplementary Documentation and Publication Policy

*Final Report:* All reporting will be performed by IPRC. The final report will address all aspects of the study and will include the interpretation of all relevant data and any conclusions from them<sup>16</sup>. A copy from the final report shall be reserved by IPRC after the completion the study. A sample informed consent form, a sample CRF, a copy of the IRB approval, the bioanalytical report including method validation report and 20% chromatograms will be appended to the final report. The subjects' CRFs, clinical laboratory tests, standard calibration curves and quality control samples shall be supplemented on request. The final report shall be signed by the IPRC Investigator(s) and submitted to the sponsor with the other study supplements<sup>17</sup>.

Source Documents: Source documents include original documents, data, and records (e.g., hospital records, clinical and office charts, laboratory notes, memoranda, accountability records, recorded data from automated instruments, informed consent forms, case report forms, bioanalytical results and chromatograms, pharmacokinetic spreadsheets, copies or transcriptions certified after verification as being accurate copies, microfiches, photographic negatives, microfilms or magnetic media, x-rays, subject files, and records kept at any department involved in the trial). All Source Documents generated in connection with this study will be retained in the limited access file storage area of IPRC, respecting the privacy and confidentiality of all records that could identify the subjects. Direct access is allowed only for authorized people for monitoring and auditing purposes. Source documents shall be handled, stored and archived according to in-house procedures to assure for accurate reporting, interpretation and verification, under the supervision of the QU.

**Publication Policy:** All information concerning Test product and the Sponsor operations, such as patent applications, formulae, manufacturing processes, basic scientific data or formulation information, supplied by Sponsor and not previously published is considered confidential by the Principal Investigator and the Study Director. The results of this study are UNITHER Pharmaceuticals proprietary and cannot be published or presented in any scientific meeting without any agreement from the sponsor.





#### 9. Reference

- 1 https://www.rxlist.com/qdolo-drug.htm
- SmPC of Contramal® (100 mg/mL Oral Solution)-English Translation, date of revision of text: 04/06/2020
- "Declaration of Helsinki." As amended by the 64<sup>th</sup> WMA General assembly, Brazil, October 2013

Available at: http://www.wma.net

Guidance on Good Clinical Practice (CPMP/ICH/135/95), ICH Topic E 6 (R2), the European Medicines Agency (EMA), June 2017.

Available at:

http://www.ema.europa.eu/docs/en GB/document library/Scientific guideline/2009/09/WC 500002874.pdf

- Jordan Law for Clinical Study Conduction, 2011.
- Guidelines for the conduct of Research involving Human subjects at the National Institutes of Health. Office of Human Subjects Research (OHRP), Title 45, Part 46 Protection Of Human Subjects

Available at: http://www.hhs.gov/ohrp/humansubjects/guidance/45cfr46.html.

Guidance for Industry: Bioavailability and Bioequivalence Studies Submitted in NDAs or INDs — General Considerations. U.S. Department of Health and Human Services Food and Drug Administration Center for Drug Evaluation and Research (CDER), March 2014.

#### Available at:

 $\underline{https://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm389370.pdf}$ 

Guideline On The Investigation Of Bioequivalence. Committee For Medicinal Products For Human Use (CHMP), European Medicines Agency (EMA), Doc. Ref.: CPMP/EWP/QWP/1401/98 Rev. 1/ Corr, London, 20 January 2010.





Available at: <a href="http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline">http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline</a> /2010/01/WC500070039.pdf

Guidance for Industry: FDA Bioanalytical Method Validation Guidelines U.S. Department of Health and Human Services Food and Drug Administration Center for Drug Evaluation and Research (CDER) Center for Veterinary Medicine (CVM), May 2018

Available at: <a href="https://www.fda.gov/files/drugs/published/Bioanalytical-Method-Validation-Guidance-for-Industry.pdf">https://www.fda.gov/files/drugs/published/Bioanalytical-Method-Validation-Guidance-for-Industry.pdf</a>

The European Medicines Agency (EMA). Guideline on bioanalytical method validation, EMEA/CHMP/EWP/192217/2009, Committee for Medicinal Products for Human Use (CHMP), 1 February 2012.

Available at:

http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2011/08/WC 500109686.pdf

Note for Guidance on Clinical Safety Data Management; Definitions and Standards for Expedited Reporting (CPMP/ICH/377/95), ICH Topic E 2 A, The European Medicines Agency (EMA), June 1995.

Available at:

http://www.ema.europa.eu/docs/en GB/document library/Scientific guideline/2009/09/WC 500002749.pdf



Guidance for Industry: Statistical Approaches to Establish Bioequivalence. US Dept. of Health and Human Services, Food and Drug Administration (FDA), Centre for Drug Evaluation and Research (CDER), January, 2001.

Available at: http://www.fda.gov/downloads/Drugs/Guidances/ucm070244.pdf





Note For Guidance On Statistical Principles For Clinical Trials (CPMP/ICH/363/96), ICH Topic E 9, The European Medicines Agency (EMA). September 1998.

Available at:

http://www.ema.europa.eu/docs/en GB/document library/Scientific guideline/2009/09/WC 500002928.pdf

Note for Guidance on the Structure And Content Of Clinical Study Report (CPMP/ICH/137/95), ICH Topic E 3, The European Medicines Agency (EMA). July 1996.

#### Available at:

 $http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC 500002832.pdf$ 

<sup>17</sup> Note for Guidance on coordinating investigator signature of clinical study reports, (CPMP/EWP/2747/00), The European Medicines Agency (EMA). October 2001.

### Available at:

 $http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC 500003656.pdf$ 





# 10. PROTOCOL VERSION HISTORY AND SUMMARY OF CHANGES

| Version | Description of change | Change<br>carried<br>out on<br>pages | Reason of<br>Change |
|---|---|---|---|
| 1.0 | creation | NA | NA |









## ANNEX VI PROTOCOL ADMINISTRATIVE CHANGES

COMPARATIVE RANDOMIZED, SINGLE DOSE, TWO-WAY CROSSOVER OPEN LABEL STUDY TO DETERMINE THE BIOEQUIVALENCE OF 5 MG/ML TRAMADOL HYDROCHLORIDE ORAL SOLUTION (08P1902F0) RELATIVE TO CONTRAMAL® 100 MG/ML ORAL SOLUTION AFTER AN ORAL ADMINISTRATION TO HEALTHY ADULTS UNDER FASTING CONDITIONS